CLINICAL TRIAL: NCT01972399
Title: Influence of Laser Therapy Upon Surgical Treatment of Peri-implantitis Lesions.
Brief Title: Laser Therapy Treatment of Peri-implantitis.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn from IRB at PI's request
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dr Hom-Lay Wang, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00077816
Record Dates: First submitted 2013-10-07; First posted 2013-10-30 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser (Experimental): A laser will be used to clean out the area around the diseased implant to try to regain bone.
  Interventions: Procedure: Laser
- Mechanical (Active Comparator): Mechanical debridement will be used to clean out the area around the diseased implant to try to regain bone.
  Interventions: Procedure: Mechanical debridement

INTERVENTIONS:
Procedure: Laser — This is a surgery that the patient will undergo and the laser will be used to clean the surface of the implant.
  Arms: Laser
Procedure: Mechanical debridement — This is a surgery that the patient will undergo to have the surface of the implant cleaned using hand instruments.
  Arms: Mechanical

SUMMARY:
The primary objective of this study is to compare the clinical outcomes of using Er: YAG laser along with bone graft and barrier membrane to conventional mechanical debridement also with bone graft and barrier membrane in the treatment of peri-implantitis infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 18 - 85 years
* Physical status according to the American Society of Anesthesiologists (ASA) I or II, which includes patients who are systemically healthy or suffer under mild to moderate, but well controlled systemic diseases.
* Patients having a minimum of 1 dental implant with peri-implantitis.
* The dental implant with peri-implantitis has ≥ 3 threads exposed or pocket probing depth (PPD) ≥ 5mm, with bleeding on probing (BOP) and/or suppuration (pus).
* The implants are in function for at least 6 months
* No uncontrolled systemic disease or condition known to alter bone metabolism, like Osteoporosis, Osteopenia, Hyperparathyroidism, Paget's disease.
* Only rough surface implant will be included in this study

Exclusion Criteria:

* Long-term use of antibiotics > 2 weeks in the past two months
* No peri-implantitis treatment in the last 2 months
* Patients taking medications known to modify bone metabolism (such as bisphosphonates, corticosteroids, Hormone replacement therapy for menopausal women, Parathyroid hormone, Denosumab, strontium ranelate).
* Pregnant females or those planning to become pregnant.
* Patients with a history of medically diagnosed oral cancer, bisphosphonate usage, Sepsis or those having adverse outcomes to oral procedures in the past, will be excluded
* Mobility of dental implants
* History of alcoholism or drug abuse
* Current smokers or quit smoking less than 6 months
* Diseases of the immune system or any medical condition that may influence the outcome (uncontrolled diabetes (HbA1c >7)
* Patients with allergies known to affect one or more of the treatment provided in this study
* Polish surface implants
* Implants with trabecular surface

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Perio Probing Depth | Change in probing depth from beginning of study to 6 months after intervention

SECONDARY OUTCOMES:
Bleeding on Probing | Change in bleeding on probing from beginning of study to 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Suarez, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States